CLINICAL TRIAL: NCT05679297
Title: Structural and Functional Grey and White Matter Changes in Patients With Pain Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: European Pain Federation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-00028; ko22Papadopoulou
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Central Post-stroke Pain
Keywords: thalamic pain; thalamic stroke; chronic pain; sensory abnormalities; pain disorder; migraine
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Migraine Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with thalamic CPSP (central post-stroke pain): Patients with CPSP of thalamic origin due to stroke.
  Interventions: Diagnostic Test: Quantitative sensory testing (QST); Diagnostic Test: Magnetic resonance imaging (MRI); Other: Clinical interview/exam; Other: Follow-up interview
- Patients with thalamic stroke without CPSP: Patients with thalamic stroke at least 2 years ago, but without CPSP or other chronic pain disorders
  Interventions: Diagnostic Test: Quantitative sensory testing (QST); Diagnostic Test: Magnetic resonance imaging (MRI); Other: Clinical interview/exam; Other: Follow-up interview
- Patients with migraine: Patients with migraine (other central pain disorder)
  Interventions: Diagnostic Test: Quantitative sensory testing (QST); Diagnostic Test: Magnetic resonance imaging (MRI); Other: Clinical interview/exam
- Healthy controls: Age- and gender-matched healthy control subjects
  Interventions: Diagnostic Test: Quantitative sensory testing (QST); Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Quantitative sensory testing (QST) — The QST is a standardized, internationally accepted test battery consisting of several well-established, non-invasive tests, measuring parameters, which reflect nearly all aspects of somatosensation.
  1. Thermal detection threshold for the perception of cold, warm and paradoxical heat sensations
  2. Thermal pain threshold
  3. Mechanical detection thresholds for touch
  4. Mechanical pain threshold for pinprick stimuli
  5. Stimulus-response functions
  6. Wind- up ratio: The wind- up ratio represents the quotient of the pain intensity evoked by 10 pin-prick stimuli and the pain intensity evoked by one single pin-prick stimulus
  7. Vibration detection threshold
  8. Pressure pain threshold
Diagnostic Test: Magnetic resonance imaging (MRI) — Functional and structural MRI data will be collected using a 3 Tesla Siemens Scanner with a multi-channel head coil.
  For the resting state functional MRI the subjects will merely lie in the scanner for about 10 minutes.
  A "painful heat/cold stimulation" will be performed to study the differences in pain processing between the three groups
Other: Clinical interview/exam — The pain characteristics will be assessed through a standardized questionnaire. The german pain questionnaire is a validated questionnaire that assesses various dimensions of pain. Patients will also get a complete neurological examination by an experienced clinician.
  Groups: Patients with migraine; Patients with thalamic CPSP (central post-stroke pain); Patients with thalamic stroke without CPSP
Other: Follow-up interview — Structured telephone interview with 3 Questionnaires
  1. The german pain questionnaire
  2. Questionnaire regarding clinical development since the last visit designed by the investigators
  3. German translation of 12-item-allodynia symptom checklist (ASC-12)
  Groups: Patients with thalamic CPSP (central post-stroke pain); Patients with thalamic stroke without CPSP

SUMMARY:
The goal of this observational study is to examine the association between exact lesion location and presence of thalamic CPSP (Central post-stroke pain) in a larger number of patients after thalamic stroke.

DETAILED DESCRIPTION:
The researchers will explore how the brain areas and mechanisms of brain plasticity are involved in the generation of thalamic CPSP, compared to other pain disorders, using structural and functional magnetic resonance imaging (MRI) at 3 Tesla. The functional magnetic resonance imaging (fMRI) will be also used to assess the cerebral processing of heat/cold stimuli in patients with thalamic pain compared to thalamic stroke patients without pain, to patients with migraine (other central pain disorder) and to normal controls. In addition the researchers want to assess the somatosensory profile of thalamic pain patients and compare it with thalamic stroke patients without pain, patients with migraine (pain control) and normal controls.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thalamic central post-stroke pain (CPSP) :

   Patients fulfilling all of the following inclusion criteria are eligible for the study:
   * Informed Consent as documented by signature (Appendix Informed Consent Form)
   * History of thalamic stroke (infarction or bleed)
   * Diagnosis of definite central-post stroke pain (according to the criteria proposed by Klit et al, 2009)
   * No other chronic pain condition
   * Age: ≥18 years old
2. Patients with thalamic stroke without CPSP:

   Patients fulfilling all of the following inclusion criteria are eligible for the study:
   * Informed Consent as documented by signature (Appendix Informed Consent Form)
   * History of thalamic stroke (infarction or bleed), at least 2 years ago
   * No chronic pain condition (neither CPSP or other pain condition)
   * Age ≥18 years old
3. Patients with migraine (other pain condition):

   Patients fulfilling all of the following inclusion criteria are eligible for the study:
   * Informed Consent as documented by signature (Appendix Informed Consent Form)
   * History of highly frequent (≥8 monthly migraine days) or chronic migraine (≥15 monthly migraine days).
   * No history of stroke
   * Age ≥18 years old
4. Healthy controls:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* No history of stroke
* No chronic pain condition
* Age: ≥18 years old

Exclusion Criteria:

* History of severe neurological, internistic or psychiatric disease
* MRI related exclusion criteria:

  * paramagnetic and/or superparamagnetic foreign objects in the body (especially when located close to the brain)
  * Pacemaker
  * Claustrophobia
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment of patients with thalamic pain will take place at the Department of Neurology, University Hospital Basel in collaboration with the chronic pain service of the Department of Anesthesiology, University Hospital Basel and the "Schmerzklinik Kirschgarten" in Basel. The recruitment of patients with thalamic stroke without pain as well as of patients with migraine (other pain disorder) will take place at the Department of Neurology, University Hospital Basel, the latter especially from the "Kopfsprechstunde". Healthy subjects will be recruited by public announcements on the University Hospital's and the University's notice board and website.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
The exact lesion location in the thalamus in patients with thalamic pain compared to patients with thalamic stroke without pain | One time assessment with a duration of max. 90 minutes.
  To determine the mutual lesion location in patients with CPSP of thalamic origin in standard stereotactic space using high-resolution 3 T MRI data and to calculate odds ratio maps for the risk of developing CPSP of thalamic origin with lesion of specific areas of the thalamus.

SECONDARY OUTCOMES:
Structural gray matter changes in patients with thalamic pain compared to the other patient groups and the healthy controls | One time assessment with a duration of max. 90 minutes.
  The 3 dimensional MPRAGE images will be used to assess cortical thickness and subcortical morphometry
Structural white matter changes in patients with thalamic pain compared to the other patient groups and the healthy controls | One time assessment with a duration of max. 90 minutes.
  Diffusion Tensor Imaging (DTI) will be used to asess the integrity of the white matter
Functional brain changes regarding the connectivity of pain networks in patients with thalamic pain compared to the other patient groups and the healthy controls | One time assessment with a duration of max. 90 minutes.
  Resting state fMRI (functional MRI) will be used to assess the functional connectivity between the thalamus and cortical areas next to the default-mode network and the sensory-motor network.
Functional brain changes regarding the central processing of heat/cold stimulation in patients with thalamic pain compared to the other patient groups and the healthy controls | One time assessment with a duration of max. 90 minutes.
  Painful heat- and cold stimulation will be performed during the fMRI session at one time-point to assess the central processing of pain in all participants
Somatosensory profile of patients with thalamic pain vs. migraine (pain-control-group) | One time assessment with a duration of max. 60 minutes.
  Somatosensory profile will be assessed by quantitative sensory testing (QST). This standardized, internationally accepted test battery consists of well-established, non-invasive tests, which are performed on the face, hand or foot of the participants. The tests measure parameters which reflect nearly all aspects of somatosensation (thermal detection thresholds, thermal pain thresholds, mechanical detection thresholds for touch, mechanical pain threshold, mechanical allodynia, vibration detection threshold and pressure pain threshold).

OTHER OUTCOMES:
Assessment of severity and characteristics of pain. | Two time assessment at baseline and 8-year-follow-up with a duration of max. 60 minutes.
  Pain characteristics will be assessed by the German pain questionnaire ("Deutscher Schmerzfragebogen"). It is a detailed questionnaire for the standardized collection of relevant pain characteristics, which is commonly used in the German language area. The first 8 items (sensory adjectives) represent a qualitative sensory description of pain that can provide information for the differential diagnosis of individual pain syndromes (e.g. headache, neuropathic pain). A summary evaluation is carried out for the affective scale. For this purpose, the total value (0-12) is formed from the individual ratings (each from 0 to 3) of the last four items (affective adjectives: miserable, horrid, horrible, terrible). A total value of 8 (corresponds to a percentage of 75%) can be set as the limit value for an increased affective experience of pain; values above this are to be assessed as conspicuous.
Longitudinal evaluation of clinical development in CPSP | One time assessment with a duration of max. 10 minutes.
  The clinical development of CPSP will be assessed by an 8-year follow-up interview via phone call. The interview/questionnaire consists of 6 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Athina Papadopoulou, PD Dr. med., Principal Investigator — University Hospital Basel, Department of Neurology
Locations (1):
- University Hospital Basel, Department of Neurology, Basel, Switzerland